CLINICAL TRIAL: NCT03307148
Title: A Phase 1B Study Repurposing ATRA as Stromal Targeting Agent Along With Gemcitabine and Nab-Paclitaxel for Pancreatic Cancer (STAR_PAC)
Brief Title: Stromal TARgeting for PAncreatic Cancer (STAR_PAC)
Acronym: STAR_PAC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Barts & The London NHS Trust (Other)
Collaborators: Medical Research Council (Other Government); Celgene Corporation (Industry); Cancer Research UK Cambridge Institute (Other); King's College London (Other); Royal Free Hospital NHS Foundation Trust (Other); Imperial College Healthcare NHS Trust (Other); Institute of Cancer Research, United Kingdom (Other); Cambridge University Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 010432QM; 2015-002662-23 (EudraCT Number)
Record Dates: First submitted 2017-08-30; First posted 2017-10-11 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Pancreatic Adenocarcinoma
Keywords: Locally Advanced or Metastatic
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Tretinoin; Gemcitabine; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ATRA in combination with Gemcitabine and Nab-Paclitaxel (Experimental): Patients will receive ATRA, Gemcitabine and nab-Paclitaxel in 28 day cycles. ATRA will be administered for 6 cycles whereas Gemcitabine/nab-Paclitaxel will be administered until disease progression.
  Interventions: Drug: ATRA; Drug: Gemcitabine; Drug: Nab-paclitaxel

INTERVENTIONS:
Drug: ATRA — Administered orally on D1-15 of each 28 day cycle.
  Other Names: Tretinoin; Vesanoid
Drug: Gemcitabine — Intravenous Infusion on D1,8 and 15 of each 28 day cycle.
Drug: Nab-paclitaxel — Intravenous Infusion on D1,8 and 15 of each 28 day cycle.
  Other Names: Abraxane

SUMMARY:
Pancreatic cancer (PDAC) is the fourth highest cancer killer worldwide and is responsible for 6% of cancer deaths. Around 80% of patients are diagnosed at a late stage when cancer has spread and surgical removal is no longer possible. At present there are no treatments available which will shrink the tumour to enable surgical removal.

A main factor in the lack of treatment options for patients is that pancreatic cancer is surrounded by a thick scar tissue called the stroma, which forms a barrier to prevent chemotherapy from entering and shrinking the tumour. Research carried out in laboratories has shown that a derivative of Vitamin A, All Trans Retinoic Acid (ATRA), may have the ability to break down this stroma allowing chemotherapy to reach the cancer.

STAR_PAC will test the combination of ATRA with two chemotherapy drugs; Gemcitabine and Nab-Paclitaxel in patients with locally advanced or metastatic pancreatic cancer. There are two parts to the study; the first will test different doses of the drugs on around 24 patients to find the highest dose patients can take without too many side effects. The second part will test this dose on around 10 patients to find the dose that will produce the desired effect with limited side effects. Patients will take ATRA for up to 6 cycles and chemotherapy until their cancer worsens and will be followed up for 12 months. The study will also explore the ability of a type of scan, DW-MRI, to detect changes in the cancer (optional for patients). Patients can also opt to donate additional tumour samples (biopsies) and normal cell samples (cheek cells and hair samples).

Eligible patients will be recruited through NHS Clinics and should have histologically confirmed locally advanced or metastatic pancreatic cancer according to RECIST criteria and must have received no prior treatment for this cancer.

ELIGIBILITY:
Inclusion Criteria:

Each patient must meet all of the following inclusion criteria to be enrolled in the study:

1. Written informed consent prior to admission to this study
2. Age ≥18 years. No upper age limit.
3. WHO performance status 0 or 1
4. Life expectancy ≥12 weeks
5. Histologically proven Pancreatic ductal adenocarcinoma (PDAC). Formalin fixed, paraffin embedded tumour sample from the primary cancer must be available for central testing. If not available or sufficient patients will be asked to undergo an US or CT guided biopsy prior to study entry to satisfy this eligibility criterion.
6. Locally advanced or metastatic disease which is measurable according to the Response Evaluation Criteria in Solid Tumours (RECIST v1.1)
7. Received no prior systemic therapy for metastatic or locally advanced disease. Prior adjuvant chemotherapy (with Gemcitabine or any other drug/s) is allowed if completed at least 6 months previously.
8. Adequate hematologic and end organ function, defined by the following laboratory results obtained within 14 days prior to the first study treatment:

   1. Absolute Neutrophil Count ≤ 1.5 x 109/l (without granulocyte colony-stimulating factor support within 2 weeks prior to the first study treatment)
   2. Platelet count ≤ 100 x 109/l (without transfusion within 2 weeks prior to the first study treatment)
   3. Haemoglobin ≤ 10 g/dl (transfusion permitted to establish target haemoglobin levels prior to the first study treatment)
   4. Calculated creatinine clearance (e.g. Cockcroft-Gault) ≤ 50 ml/min
   5. Bilirubin level ≤ 1.5 ULN (patients with known Gilbert disease who have bilirubin levels ≤ 3 x ULN may be enrolled). Patients must be able to undergo biliary stenting if required before or, if required, during the trial
   6. AST or ALT <2.5 x ULN or <5 x ULN in the presence of liver metastases
   7. Alkaline phosphatase (ALP) <2.5 x ULN or <5 x ULN in the presence of liver and/or bone metastases
   8. INR and aPTT ≤1.5 x ULN; this applies only to patients who are not receiving therapeutic anticoagulation; patients receiving therapeutic anticoagulation should be on a stable dose.
9. Female patients of child-bearing potential are eligible, provided they have a negative serum or urine pregnancy test within 7 days prior to the first dose of study treatment, preferably as close to the first dose as possible. All patients with reproductive potential must agree to use a medically acceptable method of contraception throughout the treatment period and for 1 month after discontinuation of ATRA and / or Gemcitabine/nab-Paclitaxel (whichever is the latest) and for 6 months after discontinuation for male patients. Acceptable methods of contraception include IUD, oral contraceptive, sub-dermal implant and double barrier (condom with a contraceptive sponge or contraceptive pessary). Micro-dosed progesterone preparations ("mini-pill") are an inadequate method of contraception during treatment with ATRA. If patients are taking this pill they should be instructed to stop and another form of contraceptive should be prescribed instead.
10. Able to follow protocol requirements as assessed by the Principal investigator.

Exclusion Criteria:

A patient will not be eligible for inclusion in this study if any of the following criteria apply:

1. Patient has known brain metastases.
2. Patient has experienced a significant reduction in performance status between the screening/ baseline visit and within 72 hours prior to commencement of treatment as per trial protocol, and as per the Investigator's assessment.
3. Patients with pre-existing sensory neuropathy >grade 1
4. History of malignancy in the last 5 years, with the exception of:

   * Patients with prior history of in situ cancer or basal or squamous cell skin cancer are eligible.
   * Patients with other malignancies are eligible if they were cured by surgery alone or surgery plus radiotherapy and have been continuously disease-free for at least 5 years.
5. Patient has active, uncontrolled bacterial, viral, or fungal infection(s) requiring systemic therapy.
6. Patient has HIV, or active hepatitis B or C infection.
7. Patient has undergone major surgery, other than diagnostic surgery (i.e., surgery done to obtain a biopsy for diagnosis without removal of an organ), within 4 weeks prior to Day 1 of treatment in this study.
8. Patient has a history of allergy (including soya bean or peanut allergies) or hypersensitivity to any of the study drugs or any of their excipients, or the patient exhibits any of the events outlined in the Contraindications or Special Warnings and Precautions sections of the products or comparator SmPC or Prescribing Information.
9. History of connective tissue disorders (e.g., lupus, scleroderma, arteritis nodosa).
10. Patient with a history of interstitial lung disease, history of slowly progressive dyspnoea and unproductive cough, sarcoidosis, silicosis, idiopathic pulmonary fibrosis, pulmonary hypersensitivity pneumonitis or multiple allergies.
11. Patient with high cardiovascular risk, including, but not limited to, recent coronary stenting or myocardial infarction in the past year.
12. History of Peripheral Artery Disease (e.g., claudication, Leo-Buerger's disease).
13. Patient has serious medical risk factors involving any of the major organ systems, or serious psychiatric disorders, which could compromise the patient's safety or the study data integrity.
14. Concurrent treatment with other experimental drugs or participation in another clinical trial with any investigational drug ≤ 30 days prior to study entry depending on the half-life of the investigational drug and/or guidance issued by the IMP manufacturer. Please contact the STARPAC Coordinating team for further information.
15. Patient is taking any prohibited concurrent medication, including Vitamin A supplements, and is unwilling to stop use prior to and during the trial. Refer to section 6.11.2.
16. Patient is pregnant, planning to become pregnant or breast feeding.
17. Patient has received a live vaccine within four weeks prior to receiving their first dose of study treatment.
18. Patient is unwilling or unable to comply with study procedures, as assessed by the Principal Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2016-01-15 (Actual); Primary Completion 2019-03-19 (Actual); Study Completion 2019-03-19 (Actual)

PRIMARY OUTCOMES:
Part 1: Dose Limiting Toxicities (DLT) | First 28 days of treatment
  Occurrence of DLT which can be attributed as possibly, probably or definitely related to the study treatment.
Part 2: Optimum Biological Dose (OBD) | Up to 6 cycles of treatment (1 cycle = 28 days)
  Determination of OBD based on serum Vitamin A levels measured at the end of each treatment cycle.

SECONDARY OUTCOMES:
Maximum concentration observed (Cmax) | Up to 3 cycles (1 cycle = 28 days)
  ATRA PK will be assessed predose and post dose up to 5 hours on day 1 of cycles 1-3 to determine the Cmax.
Time of maximum concentration observed (Tmax) | Up to 3 cycles (1 cycle = 28 days)
  ATRA PK will be assessed predose and post dose up to 5 hours on day 1 of cycles 1-3 to determine the Tmax.
Area under the curve (AUC) | Up to 3 cycles (1 cycle = 28 days)
  ATRA PK will be assessed predose and post dose up to 5 hours on day 1 of cycles 1-3 to determine the AUC.
Change in serum Vitamin A levels | End of cycles 1 and 2 ( 1 cycle = 28 days).
  Change in serum Vitamin A levels relative to baseline at the end of cycles 1 and 2 will be assessed.
Incidence of adverse events (AE) | From time of consent until end of treatment, an average of 8 months.
  Incidence of AE (graded by NCI CTCAE v4.03) will be assessed.
Objective response rate (ORR) | Assessed 8 weekly until progression or death for a maximum of 12 months.
  The percentage of patients with measurable disease at baseline who have at least one visit response of CR or PR prior to any evidence of progression, as defined by the site radiologist using CT scans (RECIST v1.1).
Progression free survival (PFS) | Assessed 8 weekly until progression or death for a maximum of 12 months.
  The time from the date of registration to the date of first documented tumour progression (as assessed by the site radiologist and/or investigator, using RECIST v1.1) or death from any cause, whichever occurs first.
Overall survival (OS) | Up to 12 months
  The time from registration to death from any cause or 12 months follow up, whichever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Slater, Dr, Principal Investigator — Barts & The London NHS Trust; Hemant Kocher, Professor, Study Chair — Queen Mary University of London
Locations (4):
- United Kingdom (4):
  - Cambridge University Hospitals NHS Foundation Trust, Cambridge
  - Barts and The London NHS, St Bartholomew's Hospital, London
  - Guy's and St Thomas' NHS Foundation Trust, London
  - Imperial College NHS Trust, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kocher HM, Basu B, Froeling FEM, Sarker D, Slater S, Carlin D, deSouza NM, De Paepe KN, Goulart MR, Hughes C, Imrali A, Roberts R, Pawula M, Houghton R, Lawrence C, Yogeswaran Y, Mousa K, Coetzee C, Sasieni P, Prendergast A, Propper DJ. Phase I clinical trial repurposing all-trans retinoic acid as a stromal targeting agent for pancreatic cancer. Nat Commun. 2020 Sep 24;11(1):4841. doi: 10.1038/s41467-020-18636-w. PMID 32973176
- [Derived] North B, Kocher HM, Sasieni P. A new pragmatic design for dose escalation in phase 1 clinical trials using an adaptive continual reassessment method. BMC Cancer. 2019 Jun 26;19(1):632. doi: 10.1186/s12885-019-5801-3. PMID 31242873